CLINICAL TRIAL: NCT02056184
Title: Targeted Ultrasound in Rheumatoid Arthritis
Acronym: TURA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: AbbVie (Industry); Theorem (Unknown)
Responsible Party: Principal Investigator, Paul Emery, Chief Investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HG/1096; RR13/10787 (Other: Sponsor reference); 2013-002777-22 (EudraCT Number)
Record Dates: First submitted 2014-01-30; First posted 2014-02-05 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Rheumatoid Arthritis; Targeted Ultrasound
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adalimumab, masked ultrasound (Active Comparator): Adalimumab and blinded ultrasound.
  Interventions: Drug: Adalimumab
- Adalimumab, unmasked ultrasound (Experimental): Adalimumab and open ultrasound.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab
  Other Names: Humira

SUMMARY:
The purpose of this study is to determine whether therapy modifications (including addition of ultrasound-guided treatment change) can change imaging results in patients with early rheumatoid arthritis in a stable clinical disease activity state.

DETAILED DESCRIPTION:
Rheumatoid arthritis is the most common form of inflammatory arthritis. It is a condition where the body's joints become swollen and damaged. Currently, the approach used to manage rheumatoid arthritis is the so-called 'Treat to Target' approach. The aim of this approach to treatment is to achieve the absence of signs and symptoms, or best possible state of low disease activity. It requires the use of frequent routine clinical assessments to help determine what treatment to use. Ultrasound imaging (using sound waves to take images of the joints and surrounding tissues) has been shown to be better than standard clinical measurements in detecting disease activity. Doctors are already using ultrasound imaging as part of their decisionmaking, in terms of diagnosis and altering treatments, but it is has not been clearly shown if this is associated with a better control of the disease.

Participants will be randomly put into 1 of 2 treatment groups (standard treatment group or the imaging group). All patients will also undergo the ultrasound assessment. In the standard treatment arm, the doctor will not know the ultrasound result and will base treatment on the routine disease activity score alone. In the imaging group, doctors will use routine clinical disease activity score plus the ultrasound result to make decisions on which treatment is given and treatment will be increased if necessary. However, for patients in the imaging group, even if their rheumatoid arthritis remains stable as judged by the disease activity score, treatment will be increased based on signs of active disease on the ultrasound.

Participation will last for 2 years. During the study participants will be required to attend 8 clinic visits. Approximately 400 patients from a number of countries in Europe and Japan are expected to take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Confirmed Participation by Informed Consent
* Patients fulfilling the ACR/EULAR classification criteria 2010 for rheumatoid arthritis (RA)

Patients must be:

* Within the first year of starting on methotrexate AND
* Within 5 years of diagnosis AND
* In a stable clinical disease activity state (clinical remission/LDAS /other physician deemed state) on methotrexate (as monotherapy or combination +/≤ prednisolone 5mg oral daily) for at least 8 successive weeks (with no change in Disease-Modifying Anti-Rheumatic Drugs (DMARD) +/steroid therapy - see exclusion criteria)
* Female subjects must be either postmenopausal for at least 1 year, surgically incapable of childbearing, or effectively practicing an acceptable method of contraception (oral/parenteral /implantable hormonal contraceptives, intrauterine device or barrier and spermicide). Subjects must agree to use adequate contraception during the study and for at least 5 months after study completion (or longer if on relevant therapy and in line with local regulations).
* Male subjects must agree to ensure they or their female partner(s) use adequate contraception during the study and for at least 5 months after the end of the study period.

Exclusion Criteria

* Patients not on a stable dose of methotrexate within 8 weeks of screening, intolerance or contraindications (as per clinician judgment)
* Intramuscular, intraarticular or change in oral corticosteroid within 8 weeks of screening visit.
* Oral Prednisolone dose > 5 mg within 8 weeks of screening
* Treatment with any investigational agent within 4 weeks (or 5 halflives of the investigational drug, whichever is longer) of screening.
* Patients who have previously received any biological therapy for RA.
* History of severe allergic or anaphylactic reactions to human, humanised or murine monoclonal antibodies
* Evidence of serious +/uncontrolled concomitant disease which in the investigator's judgment would deem the patient inappropriate for inclusion in the study: including (but not exclusively)including cardiovascular (NYHA class III/IV heart failure), nervous system (demyelination), pulmonary (including obstructive pulmonary disease, pulmonary fibrosis), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, or Crohn's disease.).
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds).
* Any major episode of infection requiring hospitalisation or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening. Patients with persistent infections and patients at significant risk of infection (e.g. leg ulceration, indwelling urinary catheter, septic joint within 1 year (or ever if prosthetic joint still in situ).
* Active TB requiring treatment within the previous 3 years. Patients should be screened for latent TB (as per local guidelines) and, if positive, treated following local practice guidelines prior to commencing the study. Patients previously treated for tuberculosis with no recurrence in 3 years are permitted.
* Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation.

  12. Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (including haematological malignancies and solid tumours, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured), or breast cancer diagnosed within the previous 20 years unless related to primary disease under investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in whom there is a decrease in Power Doppler (PD) at week 48 after randomisation. | Week 48

SECONDARY OUTCOMES:
Total PD score at week 48 | Week 48

OTHER OUTCOMES:
GS (Grey Scale ultrasound)) at week 48 | Week 48
X-ray scores at 48 and 96 weeks. | Weeks 48 and 96
HAQ-DI scores at 48 and 96 weeks | Weeks 48 and 96
  Disability Index questionnaire
Bone densitometry scores at weeks 48 and 96 | Weeks 48 and 96
RA-WIS score at weeks 48 and 96 | Weeks 48 and 96
  Rheumatoid Arthritis Work Instability Scale
EQ-5D score at weeks 48 and 96 | Weeks 48 and 96
  Quality of life questionnaire
Proportion of patients requiring biological therapy at 48 and 96 weeks | Weeks 48 and 96
Development of Co-Morbidity Evaluation. | Week 96
  Data collected will include total steroid exposure, number of infection events, blood pressure control.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom